CLINICAL TRIAL: NCT06001944
Title: Investigation of the Efficacy of Blood Flow Restricted Training in Lateral Elbow Tendinopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Fulya Demirhan, Clinical Researcher, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 665912
Record Dates: First submitted 2023-06-01; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Lateral Epicondylitis; Tennis Elbow; Tendonitis Elbow
Keywords: lateral elbow tendinopathy; blood flow restriction; exercise
MeSH Terms: conditions — Tennis Elbow; Motor Activity | interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant
Masking Description: Treating therapists and patient will be aware of treatment. Grip strength objective measure will be performed by a clinician blinded to the participant's treatment group. All other outcome measures are patient-reported on outcome forms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): 8 weeks, 2 days a week, a multi-model rehabilitation program is implemented.
  Interventions: Other: Multimodal rehabilitation
- Experimental group (Experimental): 8 weeks, 2 days a week, blood flow restriction during exercise will be applied in addition to the multi-model rehabilitation program. The elbow will be placed near the elbow and the patient's systolic pressure will be used to restrict the blood flow with the recommended 40%-50% occlusion for the upper extremity, and the exercise intensity will be performed 75 times at 20-30% of 1 maximum repetition, 30-15-15-15 repetition and 30 seconds rest between sets.
  Interventions: Other: Blood flow restriction

INTERVENTIONS:
Other: Blood flow restriction — The BFR training group will be given detailed information about the technique and discussed possible side effects.The American Association of Sports Physicians (ACSM) recommends that at least 65% of 1 maximum repetition, similar to high-intensity exercise, 8-12 repetitions of resistant weight lifting strength training, can be used with low loads such as 20% to 30% of the maximum 1 repetition in therapy to caste hypertrophy and strength.
  Arms: Experimental group
Other: Multimodal rehabilitation — Patients with LDT will be informed that the condition will be gradually resolved with adequate rest and time.
  Exercise Training will consist of 3 phases.The goal is to protect the injured tissue from stress during the first phase of rehabilitation during the protective phase but not to restrict its function. In this phase, the use of counterforce breys, cold application, cyriax physiotherapy, Mill's manipulation, elbow mobilization and stretching to the wrist extensors will be applied. The program will be created taking into account the principle of proximal stability for distal mobility during the reinforcement phase. The rotator manchet will be added to the program. It will be active first in the exercise and then progresses resistantly according to the condition of the patient. After distal strengthening, the dress will be transferred to stabilization exercises where flexion and extension reveal simultaneous contraction.
  Arms: Control group

SUMMARY:
The investigators believe that blood flow-restricted training can result in increased caste hypertrophy and strength without stressing the tendon in lateral elbow tendinopathy, and that changes in local metabolic activities can be effective in the process of tendon healing. The researchers' aim in the study is to investigate the effectiveness of blood flow restriction training in lateral elbow tendinopathy for 8 weeks, in addition to the 2 days a week multi-modal physiotherapy program, which will be applied by limiting blood flow by 40-50% occlusion recommended for the upper extremity using the patient's systolic pressure to the severity of 20-30% of 1 maximum repetition, 75 repetitions including 30-15-15-15 repetitions and 30 seconds rest period between sets, remaining attached to the recommended 10-15 minutes period for the top extremity.

DETAILED DESCRIPTION:
Physiotherapy is the first step in the treatment algorithm for lateral elbow tendinopathy (LET), which is characterized by pain in the lateral epicondyl of the humerus during wrist extension and which limits hand-to-hand movements such as grabbing and thinning and consequently negatively affects hand functions. Extender carpi radialis brevis (ECRB) and extender digitorum, communis (EDC) are the muscles that contribute most to the onset of symptoms. Exercise, either alone or as part of a multimodal physiotherapy program, is central to the management of many patients with LDT. Exercise in patients with chronic LDT has been shown to result in more and faster relief of pain, less use of illness, less medical consultation, and increased working capacity. In literature, loading with recommended exercises is considered necessary to re-form the tendon, while on the other hand some patients may not tolerate this loading. For rehabilitation practitioners, it is quite difficult to design optimal exercise programs that facilitate musculo-skeletal system (MSK) adaptations while also enabling biological healing and safe loading of the injured body. In these cases, there has been a search for a new method that can generate physiological benefits associated with higher intensity training with exercise at lower loads. Increasing evidence supports the use of resistance training at a reduced load along with blood flow restriction (BFR) therapy to increase hypertrophic and force responses in skeletal muscle. The American Association of Sports Physicians (ACSM) recommends that at least 65% of the 1 maximum repetition, similar to exercising at high intensity with 8-12 repetition resistant weight lifting strength training, can be used in low loads such as 20% to 30% of 1 maximum repeat in the treatment to caste hypertrophy and strength. Effects of blood flow-restricted training on muscle lithium excitement, mechanical tension, metabolic stress, systemic and local hormones, vascular endothelial growth factor (VEGF) and oxidative stress mechanisms have been. There have been no randomized controlled studies in the literature on the effectiveness of BFR training in tendinopathies. However, case studies and series of cases have been included and no contraindications of BFR have been for patients with tendinopathy. The increasing number of studies on various diseases in the literature is a proof of this.

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 65 years of age,
* Lateral tendinopathy diagnosis,
* Have scored 33 or more out of 100 on the Patient Based Tennis elbow Assessment Test (PRTEE).

Exclusion Criteria:

* Dysfunction in the shoulder, neck and/or chest area,
* Local or generalized arthritis.
* The neurological deficit.
* Radial dysfunction,
* Limitation of arm functions,
* A history of shoulder or upper extremity pathology requiring surgery or treatment;
* Venous thromboembolism
* Inflammation or other hematological disorders.
* Coronary artery disease,
* Peripheral arterial disease or hypertension (systolic/diastolic blood pressure >140 mm Hg/90 mmHg),
* To be pregnant,
* Irritation of median nerves.
* Irritation of radial nerves.
* Irritation of the ulnar nerves,
* The pain score is less than 30 mm.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-04-11 (Actual); Primary Completion 2024-04-11 (Estimated); Study Completion 2024-04-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | Evaluation should be carried out at baseline, at the end of four weeks of the treatment, at the end of eight weeks of the treatment, and at the end of four weeks of follow-up
  In the resting position, a 100 mm long line will be drawn and patients will be asked to mark the area where they express the severity of the pain on that line.
Painless Grip Strength | Evaluation should be carried out at baseline, at the end of four weeks of the treatment, at the end of eight weeks of the treatment, and at the end of four weeks of follow-up
  Average values of 3 repeated measurements with the Baseline dynamometer will be recorded while the patient is sitting upright, at shoulder adduction, at 90 degree flexion of the elbow, supported at the middle rotation of the front arm and while the wrist is in a neutral position.
Patient-rated tennis elbow evaluation (PRTEE) | Evaluation should be carried out at baseline, at the end of four weeks of the treatment, at the end of eight weeks of the treatment, and at the end of four weeks of follow-up
  It consists of two subheadings, pain and function. Function subheadings include specific activities and general activities, and each subgroup takes a value from 0 to 10. For the total score, the average of individual and general activity scores is collected with the total pain score. The result is a value between 0 and 100.

SECONDARY OUTCOMES:
SF-12 Quality of Life Questionnaire | Evaluation should be carried out at baseline, at the end of four weeks of the treatment, at the end of eight weeks of the treatment, and at the end of four weeks of follow-up
  The SF-12 consist of 12 items assesing physical and mental health and yields 2 summary scores; the mental component summary and physical component summary. Scoring is norm based with a mean of 50; higher scores indicate better health.
Global Rating of Change | Evaluation should be carried out at baseline, at the end of four weeks of the treatment, at the end of eight weeks of the treatment, and at the end of four weeks of follow-up
  Global rating of change scale quantifies a patient's improvement or deterioration over time, and identifies the effect of an intervention or charts the clinical course of a condition. The patient selects between "much worse", "slightly worse", "stayed at same", "slightly better" and, "much better".
Range of Motion | Evaluation should be carried out at baseline, at the end of four weeks of the treatment, at the end of eight weeks of the treatment, and at the end of four weeks of follow-up
  The range of motion clarity of the shoulder, elbow, front arm and wrist joints in resting position using the gonyometer will be tested.
Manual Muscle Testing | Evaluation should be carried out at baseline, at the end of four weeks of the treatment, at the end of eight weeks of the treatment, and at the end of four weeks of follow-up
  The upper, middle and lower trapezoidal muscles, serratus anterior, biceps brachii and triceps brachii will be evaluated.
Pressure-Pain Threshold Measurement | Evaluation should be carried out at baseline, at the end of four weeks of the treatment, at the end of eight weeks of the treatment, and at the end of four weeks of follow-up
  An algometer is a device consisting of a frame displaying the pressure to be applied to this piston with a metal piston containing a round disk of about 1 cm in diameter at the end. The algometer will be asked to tell the patient the level of discomfort by pressing it at a straight angle to the most sensitive area in the lateral epicondyl area. The pressure value for the pain sensation will be determined as the pain threshold and the values obtained in kilograms (kg) will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Yıldız ANALAY AKBABA, Assoc. prof., Study Chair — Istanbul University - Cerrahpasa
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Büyükçekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YJ, Wood SM, Yoon AP, Howard JC, Yang LY, Chung KC. Efficacy of Nonoperative Treatments for Lateral Epicondylitis: A Systematic Review and Meta-Analysis. Plast Reconstr Surg. 2021 Jan 1;147(1):112-125. doi: 10.1097/PRS.0000000000007440. PMID 33002980
- [Background] Lenoir H, Mares O, Carlier Y. Management of lateral epicondylitis. Orthop Traumatol Surg Res. 2019 Dec;105(8S):S241-S246. doi: 10.1016/j.otsr.2019.09.004. Epub 2019 Sep 19. PMID 31543413
- [Background] Karanasios S, Korakakis V, Moutzouri M, Xergia SA, Tsepis E, Gioftsos G. Low-Load Resistance Training With Blood Flow Restriction Is Effective for Managing Lateral Elbow Tendinopathy: A Randomized, Sham-Controlled Trial. J Orthop Sports Phys Ther. 2022 Dec;52(12):803-825. doi: 10.2519/jospt.2022.11211. Epub 2022 Sep 13. PMID 36099170
- [Background] Coombes BK, Bisset L, Vicenzino B. Management of Lateral Elbow Tendinopathy: One Size Does Not Fit All. J Orthop Sports Phys Ther. 2015 Nov;45(11):938-49. doi: 10.2519/jospt.2015.5841. Epub 2015 Sep 17. PMID 26381484
- [Background] Ozdincler AR, Baktir ZS, Mutlu EK, Kocyigit A. Chronic lateral elbow tendinopathy with a supervised graded exercise protocol. J Hand Ther. 2023 Oct-Dec;36(4):913-922. doi: 10.1016/j.jht.2022.11.005. Epub 2023 Mar 11. PMID 36914496